CLINICAL TRIAL: NCT01341886
Title: Effect of Metformin on Decrement in Levothyroxin Dose Required for Thyroid Stimulating Hormone (TSH) Suppression in Patients With Differentiated Thyroid Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mashhad University of Medical Sciences (Other)
Responsible Party: haleh rokni, endocrine research center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: METTC
Record Dates: First submitted 2011-04-18; First posted 2011-04-26 (Estimated); Last update posted 2011-04-26 (Estimated); Status verified 2011-04

CONDITIONS: Malignant Neoplasm of Thyroid Stage I; Malignant Neoplasm of Thyroid Stage II
Keywords: differentiated thyroid cancer; THS suppression; metformin
MeSH Terms: conditions — Thyroid Neoplasms | interventions — Metformin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- metformin (Active Comparator): patients who receive metformin in addition to levothyroxine
  Interventions: Drug: Metformin
- levothyroxine (Placebo Comparator): patients who receive only levothyroxine
  Interventions: Drug: Metformin

INTERVENTIONS:
Drug: Metformin — in case group metformin is added to levothyroxine and levothyroxine is decreased by 30% .in control group levothyroxine is reduced by 30% and no metformin is added to the regimen.

SUMMARY:
Differentiated thyroid cancer is the most common neoplasm of endocrine system. After surgery and radioiodine treatment, thyroid stimulating hormone (TSH) suppression is the main goal which is achieved with levothyroxine treatment. Levothyroxine causes increased thyroid hormones which can have negative impact on bone and cardiovascular system. Anecdotal reports have shown that metformin can induce TSH suppression without change in T3 and T4 concentration. The purpose of this study was to prescribe metformin as additional drug to levothyroxin in order to decrease levothyroxine dosage.

ELIGIBILITY:
Inclusion Criteria:

* papillary or follicular thyroid cancer
* stage 1 or 2 according to TNM system version 6
* surgery and radioiodine treatment
* levothyroxine suppression treatment

Exclusion Criteria:

* cardiopulmonary failure
* liver failure
* renal failure
* pregnancy
* drugs (colestyramin, sucralfate, phenobarbital, phenytoin, carbamazepin, rifampin, amiodarone, chloroquin, androgens, sertraline, frusemide, heparin)

Max Age: 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2010-04; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
TSH | 3 months

SECONDARY OUTCOMES:
freeT3,freeT4 | 3months

CONTACTS AND LOCATIONS:
Locations (1):
- Mashad University of Medical Sciences, Mashhad, Khorasan Razavi, Iran